CLINICAL TRIAL: NCT01235091
Title: Prevention of HIV and STDs in Drug Using Women
Acronym: WTW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Linda B. Cottler, Principal Investigator, Professor of Epidemiology in Psychiatry, Washington University School of medicine
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 97-0438; R01DA011622 (NIH)
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HIV; Sexually Transmitted Diseases; Substance Abuse
Keywords: HIV prevention; substance abuse; high risk behaviors; peer intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard (Other): NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing
  Interventions: Behavioral: NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing
- SI/WWE (Experimental): NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing along with Well-Woman Exam
  Interventions: Behavioral: NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing; Behavioral: Standard Intervention plus Well-Woman Exam
- SI/WWE/PD (Experimental): NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing along with Well-Woman Exam and Peer-delivered Enhanced Intervention
  Interventions: Behavioral: NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing; Behavioral: Standard Intervention plus Well-Woman Exam and Peer-Delivered Intervention

INTERVENTIONS:
Behavioral: NIDA Cooperative Agreement Standard Intervention plus HIV/STD testing — At the end of Baseline Session I, HIV pre-test counseling, per the NIDA Cooperative Agreement, was delivered, along with education about STD prevention, and biological samples were collected to test for HIV, Hepatitis C, syphilis, chlamydia and gonorrhea. At Baseline Session II, HIV post-test counseling was conducted and women were given their random group assignment.
Behavioral: Standard Intervention plus Well-Woman Exam — At the end of Baseline Session I, HIV pre-test counseling, per the NIDA Cooperative Agreement, was delivered, along with education about STD prevention, and biological samples were collected to test for HIV, Hepatitis C, syphilis, chlamydia and gonorrhea. At Baseline Session II, HIV post-test counseling was conducted and women were given their random group assignment. This group was assigned to additionally receive a well-woman examination within seven days.
  Arms: SI/WWE
Behavioral: Standard Intervention plus Well-Woman Exam and Peer-Delivered Intervention — At the end of Baseline Session I, HIV pre-test counseling, per the NIDA Cooperative Agreement, was delivered, along with education about STD prevention, and biological samples were collected to test for HIV, Hepatitis C, syphilis, chlamydia and gonorrhea. At Baseline Session II, HIV post-test counseling was conducted and women were given their random group assignment. This group was assigned to receive a well-woman exam within seven days along with four two-hour peer-delivered educational sessions, covering health and nutrition, stress and coping, substance abuse, and HIV/AIDS.
  Arms: SI/WWE/PD

SUMMARY:
Women Teaching Women (WTW) is proposed by a team of Washington University investigators who have focused on HIV prevention efforts among out-of-treatment injecting drug users (IDUs) and crack cocaine users, since 1988. Our peer-delivered prevention model was successful in reducing cocaine use among men. The investigators believe no differences were found in drug and sexual risk behaviors for women because the intervention lacked gender-specificity. Thus, the investigators propose to tailor our previous intervention to women's needs to determine the shorter and intermediate term effectiveness of a gender-specific model on reducing drug use and sexual risks. The urgency for women-focused interventions is highlighted by increasing HIV/STD rates among women nationwide. The intervention is designed to bring the HIV prevention message to women in a public health environment. The three-arm intervention, which targets out-of-treatment drug-using women, will assess the differential impact of a woman-centered standard intervention alone, the same standard intervention plus a well-woman exam, and those plus the addition of 4 educational sessions. This proposal responds to two NIDA PAs: 95-083 (Women's HIV Risk and Protective Behaviors) and 96-018 (Drug Abuse Prevention Intervention for Women and Minorities). Our risk reduction, epidemiological and technology transfer aims include:

Risk Reduction Aims:

1. Recruit out-of-treatment female drug injectors, heroin, crack/cocaine and methamphetamine users to into an intervention aimed at reducing high risk sexual and drug use behaviors. Street outreach, bars and clubs, shelters, health fairs and daycare facilities will be used to reach these vulnerable women at risk.
2. Administer a modified theory-based, peer-delivered, gender and culture-specific intervention that encourages women to reduce their high risk drug and sexual behaviors. Women will be randomly assigned to one of three peer-delivered interventions: a modified NIDA Cooperative Agreement Standard Intervention (SI), the SI + Well-Woman Exam (SI+WWE), or the SI+Well-Woman Exam + 4 Educational Sessions (SI+WWE+4ES). The Standard Intervention will be delivered by peers; the Well-Woman Examination will be conducted by a nurse practitioner; the four 2 hour educational sessions will be conducted by peer facilitators from area drug treatment programs paired with a community mental health or health professional.
3. Assess the effectiveness of the interventions in reducing drug and sexual risk at 4 and 12 months post-intervention, controlling for baseline characteristics.
4. Evaluate the relative cost-effectiveness of each intervention.

   Epidemiologic Aim:
5. Assess: a) incidence of HIV, Hepatitis B and C, syphilis, chlamydia and gonorrhea 12 months post-intervention; b) change in HIV risk and drug and alcohol use at 4 and 12 months post-intervention; c) the effect of psychopathology on behavior change at 12 months post-intervention; d) lifetime history of substance abuse and service utilization for mental and physical problems at baseline.

   Technology Transfer Aim:
6. Disseminate findings to the scientific community, practitioners and community members in formats that are appropriate, understandable, and usable in order that the best possible women-centered intervention can be developed for reducing HIV risk behaviors. The investigators propose to create a WebSite and present findings at local, national and international symposia. Manuals describing the interventions will be developed and made available to the field.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Reported sexual activity in the prior 4 months
* Recent cocaine, heroin or amphetamine use
* Reported living in the St. Louis metropolitan area

Exclusion Criteria:

* Under age 18
* No sexual activity in the prior 4 months
* No recent use of cocaine, heroin or amphetamines
* Resides outside the St. Louis metropolitan area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2000-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda B. Cottler, PhD, MPH, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Derived] Ruger JP, Abdallah AB, Luekens C, Cottler L. Cost-effectiveness of peer-delivered interventions for cocaine and alcohol abuse among women: a randomized controlled trial. PLoS One. 2012;7(3):e33594. doi: 10.1371/journal.pone.0033594. Epub 2012 Mar 20. PMID 22448255